CLINICAL TRIAL: NCT02585531
Title: Epinephrine, Dexamethasone, and Hypertonic Saline in Children With Bronchiolitis in the Hospital General Naval de Alta Especialidad. A Randomized Controlled Trial
Brief Title: Epinephrine, Dexamethasone and Hypertonic Saline in Bronchiolitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGNAE 06
Record Dates: First submitted 2015-10-13; First posted 2015-10-23 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Dexamethasone; Epinephrine; Hypertonic saline
MeSH Terms: conditions — Bronchiolitis | interventions — Epinephrine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HS3% group (Experimental): Administration of nebulized hypertonic saline for 4 days. Hypertonic Saline 3% 3 ml.
  Interventions: Drug: Epinephrine and Dexamethasone
- ED group (Active Comparator): Administration of nebulized epinephrine and dexamethasone for 4 days. Epinephrine 1:1000 solution. Dexamethasone solution 8mg/2ml.
  Interventions: Drug: Hypertonic Saline 3%

INTERVENTIONS:
Drug: Hypertonic Saline 3% — The treatment will be administered in the following order :
  First day: 3 treatments of nebulized HS 3% 3ml of treatment with interval 20 minutes Second to fourth day: One treatment of nebulized HS 3% 3ml every 24 hours .
  Other Names: HS3%
  Arms: ED group
Drug: Epinephrine and Dexamethasone — The treatment will be administered in the following order :
  First day: One treatment of nebulized dexamethasone 4mg (1ml of dexamethasone 8mg/2ml) + 3ml NS, followed by two treatments of nebulized epinephrine (3 ml of epinephrine in a 1:1000 solution per treatment) with interval 20 minutes Second to fourth day: One treatment of nebulized dexamethasone 4 mg (1ml of dexamethasone 8mg/2ml) + 3ml Normal saline 0.9%, every 24 hours.
  Other Names: ED
  Arms: HS3% group

SUMMARY:
Bronchiolitis is one of the main reasons for consultation in primary care and emergency services, as well as the leading cause of hospitalization for lower respiratory tract infection in children under two years. There is still no consensus on the medical management of the disease, in clinical practice there is wide variability in the treatment with inhaled drugs and / or oral bronchodilators, steroids, antihistamines despite the viral etiology of the disease, which results in increased morbidity and a major economic benefit for all health services.

Several studies are in relation to the management of bronchiolitis, one of which was made during 2014 in the Naval Hospital of High Specialty which included 90 participants comparing 3 treatment. The treatments administered were: dexamethasone and epinephrine (Levogira) (ED), hypertonic saline 3% (SSH 3%)and saline 0.9% ( SS 0.9%), finding that the handling of ED and SSH 3% had lower rates of hospital admissions compared to the symptomatic management of SS 0.9%. Although the superiority of SSH3% and ED in relation to the use of SS 0.9% was demonstrated, it was not possible to establish difference statistically significant between them. Why it was considered necessary to continue the study focused on determining the difference in the effectiveness of ED and SSH 3%. Therefore, the purpose of this investigation is to determine whether there is a difference between the use of dexamethasone and epinephrine versus hypertonic saline (3%).

DETAILED DESCRIPTION:
Respiratory tract infections are one of the leading causes of consultation in the Hospital General Naval de Alta Especialidad, in the emergency department and outpatient. Only in the last year (2014) shows that a total of 2690 pediatric consultations were provided in the emergency department, 1000 of them were for respiratory tract infections, constituting an approximate percentage of 37%. This figure increased over the previous year (2013) in which emergency visits corresponding 1130 290 cases consultations with boxes airways getting a percentage of 25% is given.

Due to the high incidence of lower respiratory tract infections among patients in the pediatric ward, specifically for infants under two patients; early diagnosis of acute bronchiolitis is essential to initiate proper management without falling into the overuse of drugs that have not shown adequate results.

In the last five years it has seen an increase in cases of bronchiolitis treated in both outpatient or emergency department of the Naval General Hospital. Given these data, a priority for a reason and consensus of treatment for patients with bronchiolitis.

Faced with these alarming epidemiological data both nationally and globally, it is difficult to understand that there is no consensus on the management of this entity. Although mortality is low, it represents a high cost for society and especially for health institutions, represented by a high rate of income, empirical treatments and other logistical issues.

This document intends to obtain evidence of better treatment in the population in order to establish an optimal management without spilling resources would reduce the rate of hospital admissions, first to the Naval General Hospital of High Specialty and then unify all Naval Health centers.

All this, on a solid foundation of knowledge, with the latest revisions in the interest of the subject, in order to provide the best care to every patient. Among the treatments given in this research the application of adrenaline is included, its usefulness is based on the action that causes on alpha receptors causing vasoconstriction, decreased blood flow and inflammation, responsible for the obstruction which is part of the pathophysiology of bronchiolitis. During the investigation it was decided to use it in its natural form (Levogira) because it is less expensive and the investigators can find it in an accessible at other institutions. Studies comparing its use in relation to the racemic epinephrine, show no difference. In addition to reporting a power 30 times higher in relation to the racemic epinephrine.

The study is feasible because the drugs used in this study are within the basic framework of hospital drugs, which do not involve any cost or use of additional staff for the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 2 years of age diagnosed with bronchiolitis
* Be beneficiaries Marine
* Outpatient
* Severity of Bronchiolitis mild to moderate scale according to Difficulty rating scale Respiratory (RDAI) for bronchiolitis (RDAI score 2-8).

Exclusion Criteria:

* Patients with a history of atopy
* Patients with a history of asthma in infants.
* Patients with comorbidity
* RDAI> 9 at diagnosis.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Rate of hospital admissions | 7 days after treatment
  Tracking each patient until 7 days after treatment to verify hospitalization rate.

SECONDARY OUTCOMES:
Respiration after treatment in the First Day. | 20 minutes after administration of treatment.
  Breathing frequency after the application of nebulization in the First day of treatment (breath per minute).
Heart rate after treatment in the First Day. | 20 minutes after administration of treatment.
  Heart rate after the application of nebulization in the First day of treatment (beat per minute).
Diastolic and Systolic blood pressure after treatment in the First Day. | 20 minutes after administration of treatment.
  Diastolic and Systolic blood pressure after the application of nebulization in the First day of treatment (mmHg).
Oxygen Saturation After after treatment in the First Day. | 20 minutes after administration of treatment.
  Oxygen Saturation after the application of nebulization in the First day of treatment (%).

CONTACTS AND LOCATIONS:
Overall Officials: Dra. Mayra Rubi Arcos Cruz, Pediatrician, Principal Investigator — Secretaria de Marina
Locations (1):
- Hospital General Naval de Alta Especialidad, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Nebot MS, Teruel GC, Cubells CL, Sabadell MD, Fernandez JP. [Acute bronchiolitis clinical practice guideline: recommendations for clinical practice]. An Pediatr (Barc). 2010 Oct;73(4):208.e1-10. doi: 10.1016/j.anpedi.2010.04.015. Epub 2010 Jul 14. Spanish. PMID 20634158
- [Result] Zorc JJ, Hall CB. Bronchiolitis: recent evidence on diagnosis and management. Pediatrics. 2010 Feb;125(2):342-9. doi: 10.1542/peds.2009-2092. Epub 2010 Jan 25. PMID 20100768
- [Result] Corneli HM, Zorc JJ, Holubkov R, Bregstein JS, Brown KM, Mahajan P, Kuppermann N; Bronchiolitis Study Group for the Pediatric Emergency Care Applied Research Network. Bronchiolitis: clinical characteristics associated with hospitalization and length of stay. Pediatr Emerg Care. 2012 Feb;28(2):99-103. doi: 10.1097/PEC.0b013e3182440b9b. PMID 22270499
- [Result] Vinci R, Bauchner H. Bronchiolitis, deception in research, and clinical decision making. JAMA. 2014 Aug 20;312(7):699-700. doi: 10.1001/jama.2014.8638. No abstract available. PMID 25138330
- [Result] Acosta A et all. Diagnóstico y manejo en niños con Bronquiolitis en fase aguda, México: Secretaria de Salud. Catálogo Maestro de Guías de práctica clínica IMSS-032-08. 2010.
- [Result] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Result] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Result] Koehoorn M, Karr CJ, Demers PA, Lencar C, Tamburic L, Brauer M. Descriptive epidemiological features of bronchiolitis in a population-based cohort. Pediatrics. 2008 Dec;122(6):1196-203. doi: 10.1542/peds.2007-2231. PMID 19047234
- [Result] Baraldi E, Lanari M, Manzoni P, Rossi GA, Vandini S, Rimini A, Romagnoli C, Colonna P, Biondi A, Biban P, Chiamenti G, Bernardini R, Picca M, Cappa M, Magazzu G, Catassi C, Urbino AF, Memo L, Donzelli G, Minetti C, Paravati F, Di Mauro G, Festini F, Esposito S, Corsello G. Inter-society consensus document on treatment and prevention of bronchiolitis in newborns and infants. Ital J Pediatr. 2014 Oct 24;40:65. doi: 10.1186/1824-7288-40-65. PMID 25344148
- [Result] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Result] Ochoa Sangrador C, Gonzalez de Dios J; Grupo Investigador del Proyecto aBREVIADo (BRonquiolitis-Estudio de Variabilidad, Idoneidad y ADecuacion). [Management of acute bronchiolitis in spanish emergency wards: variability and appropriateness analysis (aBREVIADo project)]. An Pediatr (Barc). 2013 Sep;79(3):167-76. doi: 10.1016/j.anpedi.2013.01.015. Epub 2013 Mar 6. Spanish. PMID 23481463
- [Result] Yusuf S, Caviness AC, Adekunle-Ojo AO. Risk factors for admission in children with bronchiolitis from pediatric emergency department observation unit. Pediatr Emerg Care. 2012 Nov;28(11):1132-5. doi: 10.1097/PEC.0b013e31827132ff. PMID 23114233
- [Result] Ipek IO, Yalcin EU, Sezer RG, Bozaykut A. The efficacy of nebulized salbutamol, hypertonic saline and salbutamol/hypertonic saline combination in moderate bronchiolitis. Pulm Pharmacol Ther. 2011 Dec;24(6):633-7. doi: 10.1016/j.pupt.2011.09.004. Epub 2011 Sep 29. PMID 21978929
- [Result] Ralston S, Garber M, Narang S, Shen M, Pate B, Pope J, Lossius M, Croland T, Bennett J, Jewell J, Krugman S, Robbins E, Nazif J, Liewehr S, Miller A, Marks M, Pappas R, Pardue J, Quinonez R, Fine BR, Ryan M. Decreasing unnecessary utilization in acute bronchiolitis care: results from the value in inpatient pediatrics network. J Hosp Med. 2013 Jan;8(1):25-30. doi: 10.1002/jhm.1982. Epub 2012 Oct 9. PMID 23047831
- [Result] Plint AC, Johnson DW, Patel H, Wiebe N, Correll R, Brant R, Mitton C, Gouin S, Bhatt M, Joubert G, Black KJ, Turner T, Whitehouse S, Klassen TP; Pediatric Emergency Research Canada (PERC). Epinephrine and dexamethasone in children with bronchiolitis. N Engl J Med. 2009 May 14;360(20):2079-89. doi: 10.1056/NEJMoa0900544. PMID 19439742
- [Result] Hartling L, Fernandes RM, Bialy L, Milne A, Johnson D, Plint A, Klassen TP, Vandermeer B. Steroids and bronchodilators for acute bronchiolitis in the first two years of life: systematic review and meta-analysis. BMJ. 2011 Apr 6;342:d1714. doi: 10.1136/bmj.d1714. PMID 21471175
- [Result] Brand PL, Baraldi E, Bisgaard H, Boner AL, Castro-Rodriguez JA, Custovic A, de Blic J, de Jongste JC, Eber E, Everard ML, Frey U, Gappa M, Garcia-Marcos L, Grigg J, Lenney W, Le Souef P, McKenzie S, Merkus PJ, Midulla F, Paton JY, Piacentini G, Pohunek P, Rossi GA, Seddon P, Silverman M, Sly PD, Stick S, Valiulis A, van Aalderen WM, Wildhaber JH, Wennergren G, Wilson N, Zivkovic Z, Bush A. Definition, assessment and treatment of wheezing disorders in preschool children: an evidence-based approach. Eur Respir J. 2008 Oct;32(4):1096-110. doi: 10.1183/09031936.00002108. PMID 18827155
- [Result] Lowell DI, Lister G, Von Koss H, McCarthy P. Wheezing in infants: the response to epinephrine. Pediatrics. 1987 Jun;79(6):939-45. PMID 3295741